CLINICAL TRIAL: NCT03329963
Title: Does Lifestyle Intervention Improve Bone Quality in Obese Older Adults?
Brief Title: Lifestyle Intervention to Improve Bone Quality
Acronym: LIMB-Q
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Biomedical Research Institute of New Mexico (Other)
Responsible Party: Principal Investigator, Dennis T. Villareal, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-40373; R01DK109950 (NIH)
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Aging; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifestyle intervention Group (Experimental): Behavioral therapy for weight loss and Exercise Training
  Interventions: Behavioral: Lifestyle Intervention
- Healthy lifestyle intervention Group (Active Comparator): Group education sessions that focus on diet exercise and social support.
  Interventions: Behavioral: Healthy Lifestyle Intervention

INTERVENTIONS:
Behavioral: Healthy Lifestyle Intervention — Participants in the this group will receive group educational sessions that focus on diet, exercise, and social support once a month throughout the study. The sessions will provide an opportunity for participants to discuss issues related to living with obesity and aging.Participants will also attend regular scheduled clinic visits for assessment of outcomes.
  Arms: Healthy lifestyle intervention Group
Behavioral: Lifestyle Intervention — The lifestyle modification will be achieved by group behavior therapy sessions designed to have older adults acquire positive weight-control skills/attitudes, and practice weight-maintenance skills.Participants will attend weekly group sessions (10-15 persons), which will last ~75-90 minutes. Visit frequency will be decreased to every 2 wks. from 6 to 12 mos. to prevent "treatment fatigue". A balanced diet will be prescribed to provide a deficit of 500-750 kcal/day from daily energy requirement.
  The exercise sessions are of ~90 min duration (~15 min warm-up of flexibility exercise, followed by ~30 min of aerobic exercise, and after a brief rest period, ~30 min of resistance training, and finally ~15 min balance exercise) conducted three times weekly supervised at our exercise facility for one year. Aerobic exercises consist of treadmill, stationary cycling, and stair climbing.
  Arms: Lifestyle intervention Group

SUMMARY:
Obese older adults will be randomized to participate in either healthy lifestyle intervention or behavioral diet and exercise intervention for one year. This study aims to determine the effects of Lifestyle intervention on bone microarchitecture, bone strength, bone material properties, and the mechanism behind it.

DETAILED DESCRIPTION:
Previous studies had suggested that lifestyle therapy (diet plus exercise) resulting in weight loss in elderly population improves physical function, cardio metabolic risk factors, and cognition/quality of life, but a major complication is loss of BMD. The addition of exercise to diet-induced weight loss attenuated but did not eliminate weight-loss-induced reduction of BMD. Moreover, while long-term maintenance of weight loss and physical function was feasible, sustained lifestyle change led to continued loss of hip BMD, which might predict hip fractures. Although similar BMD loss with weight loss has been observed in younger populations, BMD loss in older adults might be of particular concern because of aggravation of age-related bone loss. Moreover, the belief that obesity protects against fractures has now been challenged by studies demonstrating that obesity is associated with poor bone quality and ankle and leg fractures.Because of previous lack of options to assess bone quality in vivo, there has been little or no scientific study of the possibility that lifestyle therapy in obese older adults improves bone quality. This study represents an unprecedented opportunity to prove the hypothesis that lifestyle therapy intervention improves bone quality and thus, may confer a protective rather than adverse effect on bone health. This will be the first randomized controlled trial (RCT) to comprehensively assess bone quality using novel techniques in response to lifestyle therapy in obese older adults, with major ramifications with regards to defining optimal treatment strategies for this increasingly high-risk older population.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 - 85 years • BMI 30 kg/m2 or more• Stable body weight (±2 kg) during the past 6 months • Sedentary (regular exercise <1 h/wk. or <2 x/wk. for the last 6 months) • Willing to provide informed consent

Exclusion Criteria:

* Failure to provide informed consent.
* Any major chronic diseases, or any condition that would interfere with exercise or dietary restriction, in which exercise or dietary restrictions are contraindicated, or that would interfere with interpretation of results
* Cardiopulmonary disease (e.g. recent myocardial infarction, unstable angina, stroke) or unstable disease (e.g., New York Heart Class III or IV congestive heart failure, severe pulmonary disease requiring steroid pills or the use of supplemental oxygen ) that would contraindicate exercise or dietary restriction
* Severe orthopedic (e.g. awaiting joint replacement) and/or neuromuscular (e.g. multiple sclerosis, amyotrophic lateral sclerosis, active rheumatoid arthritis) disease or impairments that would contraindicate participation in exercise
* Other significant co-morbid disease that would impair ability to participate in the exercise-based intervention (e.g. renal failure on hemodialysis, severe psychiatric disorder [e.g. bipolar, schizophrenia], excess alcohol use [more than14 drinks per week])
* Severe visual or hearing impairments that would interfere with following directions
* Significant cognitive impairment, defined as a known diagnosis of dementia or positive screening test for dementia using the Mini-Mental State Exam score less than 24)
* Uncontrolled hypertension (BP>160/90 mm Hg)
* History of malignancy during the past 5 years (except non-melanoma skin cancers)
* Current use of bone acting drugs (e.g. use of estrogen, or androgen containing compound, raloxifene, calcitonin, parathyroid hormone during the past year or bisphosphonates during the last two years)
* Osteoporosis (T-score -2.5 and below on hip or spine scan) or history of fragility fractures - Diabetes mellitus requiring insulin for treatment or with a fasting blood glucose of >140 mg/dl, and/or HbA1c >8.5% (Those excluded from the study because of fasting blood glucose of >140 mg/dl or HbA1c>8.5% will be referred to their primary care provider for follow-up and appropriate treatment).
* Terminal illness with life expectancy less than 12 months, as determined by a physician
* Use of any drugs or natural products designed to induce weight loss within past three months.
* Positive exercise stress test for ischemia

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Change in cortical thickness | Change from baseline at 12 months
  Assessed by using high-resolution peripheral computed tomography (HR-pQCT)
Change in femoral bone strength | Change from baseline at 12 months
  Assessed by using finite element analyses (FEA) of quantitative computed tomography (QCT)

SECONDARY OUTCOMES:
Change in bone material strength | Change from baseline at 12 months
  Assessed by using microindentation testing
Change in lower extremity strength | Change from baseline at 12 months
  Assessed by using a Biodex dynamometer
Change in physical performance test | Change from baseline at 12 months
  assessed by using the objective physical performance test
Change in gait speed | Change from baseline at 12 months
  as measured by completing the time to walk a certain distance
Change in handgrip strength | Change from baseline at 12 months
  Measured by hydraulic hand dynamometer
Change in trabecular thickness | Change from baseline at 12 months
  Assessed by using HR-pQCT
Change in areal bone mineral density (BMD) | Change from baseline at 12 months
  Assessed by using dual-energy x-ray absorptiometry
Change in trabecular number | Change from baseline at 12 month
  Assessed by using HR-pQCT
Change in total volumetric BMD | Change from baseline at 12 months
  Assessed by using HR-pQCT
Change in cortical volumetric BMD | Change from baseline at 12 months
  Assessed by using HR-pQCT
Change in trabecular volumetric BMD | Change from baseline at 12 months
  Assessed by using HR-pQCT
Change in stiffness | Change from baseline at 12 months
  Assessed by using HR-pQCT
Change in trabecular separation | Change from baseline at 12 months
  Assessed by using HR-pQCT
Change in micro-finite element analyses strength | Change from baseline at 12 months
  Assessed by using HR-pQCT
Change in cortical porosity | Change from baseline at 12 months
  Assessed by using HR-pQCT
Change in general quality of life | Change from baseline at 12 months
  Assessed by using the Short Form-36 questionnaire
Change in obesity specific quality of life | Change from baseline at 12 months
  Assessed by using the Impact of weight on quality of life short form (IWQOL-Lite) questionnaire
Change in mood | Change from baseline at 12 months
  Assessed by using a mood scale questionnaire
Change in composite cognitive z-score | Change from baseline at 12 months
  Using cognitive instrument testing
Change in cardio metabolic risk factors | Change from baseline at 12 months
  Assessed by measuring metabolic syndrome components
Change in word list fluency | Change from baseline at 12 months
  Assessed by using cognitive instrument testing
Change in Ray Auditory verbal learning test | Change from baseline at 12 months
  Assessed by using cognitive instrument testing
Change in blood pressure | Change from baseline at 12 months
  Assessed by usingSphygmomanometer
Change in biochemical marker for bone turnover and bone metabolism | Change from baseline at 12 months
  Assessed by using enzyme linked immunosorbent assay and radioimmunoassay
Change in central volumetric BMD | Change from baseline at 12 months
  Assessed by using CT scan at the spine and hip
Change in waist circumference | Change from baseline at 12 months
  Assessed by using tape measurement
Change in lean mass | Change from baseline at 12 months
  Assessed by using dual-energy x-ray absorptiometry
Change in fat mass | Change from baseline at 12 months
  Assessed by using dual-energy x-ray absorptiometry
Change in visceral fat | Change from baseline at 12 months
  Assessed by using dual-energy x-ray absorptiometry
Change in physical activity using accelerometer | Change from baseline at 12 months
  Assessed by using an accelerometer
Change in body weight | Change from baseline at 12 months
  Assessed by using weighing scale
Change in sclerostin | Change from baseline at 12 months
  Assessed by using enzyme linked immunoassay
Change in wnt signaling pathways | Change from baseline at 12 months
  Assessed by measurements of circulating levels of Wnt 5a and Sfrp5
Change in total body mass | Change from baseline at 12 months
  Assessed byusing dual energy x-ray absorptiometry
Change in hormones | Change from baseline at 12 months
  Assessed by usingenzyme link immunoassay
Change in thigh mass | Change from baseline at 12 months
  Assessed by using CT scan
Change in circulating cytokines | Change from baseline at 12 months
  Assessed by using enzyme linked immunoassay
Change in adipocytokines | Change from baseline at 12 months
  Assessed by using enzyme linked immunoassay
Change in total volumetric BMD | Change from baseline at 12 months
  Assessed by using QCT Pro software
Change in cortical trabecular BMD | Change from baseline at 12 months
  Assessed by using QCT Pro software
Change in aerobic capacity | Change from baseline at 12 months
  Assessed by using indirect calorimetry during graded treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E Debakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gregori G, Mediwala S, Liebschner M, Kim D, Bryant MS, Klonis N, Armamento-Villareal R, Qualls C, Villareal DT. Bone quality response to lifestyle intervention in older adults with obesity (LIMB-Q trial): a randomised controlled trial. Lancet Healthy Longev. 2025 Sep;6(9):100761. doi: 10.1016/j.lanhl.2025.100761. Epub 2025 Sep 18. PMID 40976254